CLINICAL TRIAL: NCT01803464
Title: Effect of Botox and Vibration on Bone in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christopher Modlesky, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R15HD071397-01 (NIH); IRB # 115648-11 (Other: Alfred I. duPont Hospital for the Children); 1R15HD071397-01 (NIH)
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Cerebral Palsy; Muscle Spasticity
Keywords: Botox; Muscle strength
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Botox plus low-magnitude vibration (Experimental): Cerebral palsy and Botox + vibration
  Interventions: Device: Low-magnitude vibration; Drug: Botox
- Botox (Experimental): Cerebral palsy and Botox
  Interventions: Drug: Botox
- Cerebral palsy control (No Intervention): Cerebral palsy without treatment
- Typically developing control (No Intervention): Typically developing

INTERVENTIONS:
Device: Low-magnitude vibration — Children will receive a daily low-magnitude vibration treatment.
  Arms: Botox plus low-magnitude vibration
Drug: Botox — Children who are candidates to receive Botox as part of their standard of care.
  Arms: Botox; Botox plus low-magnitude vibration

SUMMARY:
Cerebral palsy (CP) is a neuromuscular disorder that affects approximately 800,000 individuals in the U.S. An estimated 70-80% of these individuals have spasticity which affects ambulation and requires management. Therefore, the treatment of spasticity is a primary goal of interventions for children with CP. One treatment widely used to reduce spasticity is Botox because of its ability to temporarily paralyze a muscle. However, no studies have determined the effect of Botox treatment on bone in humans. Also, a low magnitude vibration treatment has been shown to improve bone structure in the lower extremity bones of children with CP. The aims of this study are: 1) to determine the effect of Botox treatment in conjunction with a daily vibration treatment on bone mass and bone structure in children with spastic CP, and 2) to identify the mechanism that underlies the effect of Botox and vibration on bone.

DETAILED DESCRIPTION:
The investigators have been working with children diagnosed with cerebral palsy (CP) for the past 10 years. The investigators have found that bone structure is markedly underdeveloped and bone strength is severely compromised in children with CP. Also, an increased fracture rate has been observed in the lower extremity bones of children with CP. There is evidence that Botox, which is used to treat spasticity in CP, can improve motor function; however the effect of Botox on human bone is unknown. There is also evidence that low magnitude vibration treatment can improve bone mass and bone structure. The overall goal of this current research study is to investigate the effect and mechanism of action of Botox and vibration on bone in children with CP. The investigators will also examine the effect of Botox on muscle volume.

A total of 36 participants will participate in this study. The investigators will assess bone structure and muscle volume using MRI. The investigators will assess bone mass using dual-energy X-ray absorptiometry (DXA).

ELIGIBILITY:
Inclusion (Children with CP):

1. Have spastic CP
2. Between 2-12 years of age
3. Recommended for Botox treatment by their physician as part of their clinical care. Those who accept Botox treatment and those who do not accept Botox treatment are both eligible for the study.
4. A score of 1-4 on the gross motor function classification scale (GMFCS)

Exclusion (Children with CP):

1. Botox treatment in the lower extremities within the last year
2. Metal rods in both legs

Inclusion (Typically developing children):

1. Between 2 and 12 years of age.
2. Match a child with CP for sex, age and race.

Exclusion(Typically developing children):

1. Neurological disorder
2. Surgery in the lower extremities within the last year.
3. Chronic medication use

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Modlesky, PhD, Principal Investigator — University of Delaware; Freeman Miller, MD, Principal Investigator — Nemours/Alfred I duPont Hospital for Children
Locations (2):
- United States (2):
  - University of Delaware, Newark, Delaware
  - Alfred I. duPont Hospital for Children, Nemours, Wilmington, Delaware

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Time Frame: Within 30 days of the request.
Access Criteria: Data access requests will be reviewed by the PIs. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Johnson DL, Miller F, Subramanian P, Modlesky CM. Adipose tissue infiltration of skeletal muscle in children with cerebral palsy. J Pediatr. 2009 May;154(5):715-20. doi: 10.1016/j.jpeds.2008.10.046. Epub 2008 Dec 25. PMID 19111321
- [Background] Modlesky CM, Subramanian P, Miller F. Underdeveloped trabecular bone microarchitecture is detected in children with cerebral palsy using high-resolution magnetic resonance imaging. Osteoporos Int. 2008 Feb;19(2):169-76. doi: 10.1007/s00198-007-0433-x. Epub 2007 Oct 26. PMID 17962918
- [Background] Rubin C, Turner AS, Muller R, Mittra E, McLeod K, Lin W, Qin YX. Quantity and quality of trabecular bone in the femur are enhanced by a strongly anabolic, noninvasive mechanical intervention. J Bone Miner Res. 2002 Feb;17(2):349-57. doi: 10.1359/jbmr.2002.17.2.349. PMID 11811566
- [Background] Judex S, Boyd S, Qin YX, Turner S, Ye K, Muller R, Rubin C. Adaptations of trabecular bone to low magnitude vibrations result in more uniform stress and strain under load. Ann Biomed Eng. 2003 Jan;31(1):12-20. doi: 10.1114/1.1535414. PMID 12572652
- [Background] Wren TA, Lee DC, Hara R, Rethlefsen SA, Kay RM, Dorey FJ, Gilsanz V. Effect of high-frequency, low-magnitude vibration on bone and muscle in children with cerebral palsy. J Pediatr Orthop. 2010 Oct-Nov;30(7):732-8. doi: 10.1097/BPO.0b013e3181efbabc. PMID 20864862
- [Background] Ward K, Alsop C, Caulton J, Rubin C, Adams J, Mughal Z. Low magnitude mechanical loading is osteogenic in children with disabling conditions. J Bone Miner Res. 2004 Mar;19(3):360-9. doi: 10.1359/JBMR.040129. Epub 2004 Jan 27. PMID 15040823
- [Result] Modlesky CM, Whitney DG, Singh H, Barbe MF, Kirby JT, Miller F. Underdevelopment of trabecular bone microarchitecture in the distal femur of nonambulatory children with cerebral palsy becomes more pronounced with distance from the growth plate. Osteoporos Int. 2015 Feb;26(2):505-12. doi: 10.1007/s00198-014-2873-4. Epub 2014 Sep 9. PMID 25199575
- [Result] Modlesky CM, Whitney DG, Carter PT, Allerton BM, Kirby JT, Miller F. The pattern of trabecular bone microarchitecture in the distal femur of typically developing children and its effect on processing of magnetic resonance images. Bone. 2014 Mar;60:1-7. doi: 10.1016/j.bone.2013.11.009. Epub 2013 Nov 20. PMID 24269277
- [Derived] Singh H, Whitney DG, Knight CA, Miller F, Manal K, Kolm P, Modlesky CM. Site-Specific Transmission of a Floor-Based, High-Frequency, Low-Magnitude Vibration Stimulus in Children With Spastic Cerebral Palsy. Arch Phys Med Rehabil. 2016 Feb;97(2):218-23. doi: 10.1016/j.apmr.2015.08.434. Epub 2015 Sep 21. PMID 26392035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 children with spastic cerebral palsy eligible for botulinum toxin treatment and typically developing children were screened. 5 children did not meet the study criteria and 57 children were invited to participate in the study, of which 29 participated in the study.
Groups:
- Botox Plus Low-magnitude Vibration: Children with cerebral palsy who are recommended for and scheduled to receive Botox treatment will randomized to also receive vibration treatment. Children will be asked to stand on a vibration plate 10 minutes per day for 6 months.
  Botox plus low-magnitude vibration: Half of the children who receive Botox treatment will be randomly assigned to receive a high-frequency, low magnitude vibration treatment. The other half of the children who receive Botox treatment and are randomly assigned to the Botox-only group will be offered the vibration treatment at the end of the study.
- Botox: Children with cerebral palsy who are recommended for and scheduled to receive Botox treatment will randomized to serve as a Botox-only group.
  Botox: Children will not receive vibration treatment. Children in the Botox-only group will be offered vibration treatment at the end of the study.
- Cerebral Palsy Control: Children with cerebral palsy who are recommended for but decline Botox treatment will serve as controls.
- Typically Developing Control: Typically developing children without cerebral palsy will serve as controls.
Period: Overall Study
Arm/Group | Botox Plus Low-magnitude Vibration | Botox | Cerebral Palsy Control | Typically Developing Control
Started | 5 | 4 | 10 | 10
Completed | 4 | 4 | 6 | 10
Not Completed | 1 | 0 | 4 | 0
Not completed — Incomplete data | 0 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox Plus Low-magnitude Vibration | Botox | Cerebral Palsy Control | Typically Developing Control | Total
Number analyzed (Participants) | 5 | 4 | 10 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.73 (2.85) | 8.50 (2.65) | 7.61 (2.22) | 8.71 (1.68) | 8.13 (2.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 3 | 9
  Male | 4 | 3 | 6 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 10 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Bone Structure
Description: Change in cortical bone volume of the middle third of the tibia from baseline to 6 months, as measured by MRI.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Botox Plus Low-magnitude Vibration | Botox | Cerebral Palsy Control | Typically Developing Control
Number analyzed (Participants) | 4 | 4 | 6 | 10
percent change | 10.4 (8.6) | 7.6 (10.2) | 6.7 (4.7) | 9.0 (4.4)
Statistical Analysis 1: Comparison: Botox Plus Low-magnitude Vibration vs Cerebral Palsy Control; Test type: Other; Cohen's d = 0.59 — Cohen's d was calculated. The % change of the Botox plus low-magnitude vibration group minus the % change of the cerebral palsy control group was the numerator. The pooled Standard Deviation (SD) of the % change for the 2 groups was the denominator
Statistical Analysis 2: Comparison: Botox vs Cerebral Palsy Control; Test type: Other; Cohen's d = 0.13 — Cohen's d was calculated. The % change of the Botox group minus the % change of the cerebral palsy control group was the numerator. The pooled SD of the % change for the 2 groups was the denominator
Statistical Analysis 3: Comparison: Cerebral Palsy Control vs Typically Developing Control; Test type: Other; Cohen's d = 0.51 — Cohen's d was calculated. The % change of the typically developing control group group minus the % change of the cerebral palsy control group was the numerator. The pooled SD of the % change for the 2 groups was the denominator

2. Secondary Outcome: Muscle Volume
Description: Change in muscle volume of the midleg from baseline to 6 months, as measured by MRI
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Botox Plus Low-magnitude Vibration: Cerebral palsy and Botox plus vibration
  Low-magnitude vibration: Children will receive a daily low-magnitude vibration treatment.
  Botox: Children who are candidates to receive Botox as part of their standard of care.
Arm/Group | Botox Plus Low-magnitude Vibration | Botox | Cerebral Palsy Control | Typically Developing Control
Number analyzed (Participants) | 4 | 4 | 6 | 10
percent change | 9.5 (13.5) | 10.9 (14.2) | 5.1 (7.4) | 3.9 (10.1)
Statistical Analysis 1: Comparison: Botox Plus Low-magnitude Vibration vs Cerebral Palsy Control; Test type: Other; Cohen's d = 0.45 — Cohen's d was calculated. The % change of the Botox plus low-magnitude vibration group minus the % change of the cerebral palsy control group was the numerator. The pooled SD of the % change for the 2 groups was the denominator
Statistical Analysis 2: Comparison: Botox vs Cerebral Palsy Control; Test type: Other; Cohen's d = 0.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cerebral Palsy Control vs Typically Developing Control; Test type: Other; Cohen's d = 0.13 — Cohen's d was calculated. The % change of the typically developing group minus the % change of the cerebral palsy control group was the numerator. The pooled SD of the % change for the 2 groups was the denominator

3. Secondary Outcome: Bone Mass
Description: Change in bone mineral content in the distal femur from baseline to 6 months, as measured by dual-energy X-ray absorptiometry (DXA)
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Botox Plus Low-magnitude Vibration | Botox | Cerebral Palsy Control | Typically Developing Control
Number analyzed (Participants) | 4 | 4 | 6 | 10
percent change | 8.1 (4.3) | 3.2 (3.9) | 4.2 (2.5) | 3.1 (3.9)
Statistical Analysis 1: Comparison: Botox Plus Low-magnitude Vibration vs Cerebral Palsy Control; Test type: Other; Cohen's d = 1.2 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Botox vs Cerebral Palsy Control; Test type: Other; Cohen's d = 0.33 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cerebral Palsy Control vs Typically Developing Control; Test type: Other; Cohen's d = 0.33 — Cohen's d was calculated. The % change of the typically developing control group minus the % change of the cerebral palsy control group was the numerator. The pooled SD of the % change for the 2 groups was the denominator

ADVERSE EVENTS:
Arm/Group | Botox Plus Low-magnitude Vibration | Botox | Cerebral Palsy Control | Typically Developing Control
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox Plus Low-magnitude Vibration (N=5) | Botox (N=4) | Cerebral Palsy Control (N=10) | Typically Developing Control (N=10)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — Participants became nauseous while standing on the vibration platform during a 10 minute session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No